CLINICAL TRIAL: NCT01920802
Title: Quantitative Assessment and Comparison of Metabolic Changes in Non-psychotic Adults Taking the Antipsychotic Medications Fanapt (Iloperidone) or Zyprexa (Olanzapine) or Placebo
Brief Title: Assessment and Comparison of Metabolic Changes in Non-psychotic Adults Taking Iloperidone or Olanzapine or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6525
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Olanzapine; iloperidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- olanzapine (Experimental): 5mg BID olanzapine for up to 4 weeks
  Interventions: Drug: olanzapine
- iloperidone (Experimental): 6mg BID iloperidone up to 4 weeks
  Interventions: Drug: iloperidone
- placebo (Placebo Comparator): BID placebo up to 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: olanzapine — 5mg BID up to 4 weeks
  Other Names: Zyprexa
  Arms: olanzapine
Drug: iloperidone — 6 mg BID up to 4 weeks
  Other Names: Fanapt
  Arms: iloperidone
Drug: Placebo — BID up to 4 weeks
  Arms: placebo

SUMMARY:
The purpose of this pilot randomized clinical trial is to begin to delineate the pathophysiological changes associated with antipsychotic associated metabolic side effects. The study will be performed in 36 healthy people between the ages of 18 and 30, who have never taken an antipsychotic, will undergo baseline laboratory tests before being randomized to 5mg BID of olanzapine or 6mg BID of iloperidone or placebo to take for up to 4 weeks. The primary outcome measure will be a correlation of early changes in leptin with weight gain. We will also record changes in food intake, resting metabolic rate, oral glucose tolerance and fasting insulin and glucose levels, lipids and inflammation markers. Subjects will be followed closely to monitor for safety throughout the 4-week study and will be discontinued if there is a medically significant change in metabolic status or other antipsychotic side effects. Metabolic assessments will be performed again at the time of discontinuation or at the end of an 4-week period, and change from baseline in the two treatment groups will be compared.

DETAILED DESCRIPTION:
Study hypotheses:

1. Early changes (baseline vs day 3) in leptin will correlate with later changes in weight (at study termination.)

   1. Olanzapine will cause the greatest increase in calorie consumption from baseline on the multi-item meal compared with iloperidone or placebo.
   2. Olanzapine subjects will report the greatest frequency/quantity of eating in food diaries, and report increased preference for calorically dense foods (ie, higher fat content) compared to iloperidone or placebo.
   3. Early markers of endocrine changes caused by olanzapine will be greater than those caused by iloperidone or placebo, and these early changes will correlate with weight gain.
2. Olanzapine will have greater effects on glucose homeostasis than iloperidone or placebo, and these effects will be separate from effects on body weight and composition.

   1. Early signs of metabolic disturbance, including glucose intolerance (greater excursion on OGTT) and insulin resistance (higher plasma insulin) will precede any significant weight gain.
   2. Early evidence of glucose intolerance and/or insulin resistance will predict greater metabolic derangements with further dosing of olanzapine, as evidenced by exacerbated glucose intolerance on OGTT or higher plasma glucose/insulin levels. These effects may not necessarily parallel weight gain.
   3. Olanzapine will be associated with greater markers of inflammation than iloperidone or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-35 with no history of any Axis-I diagnosis
* Does not meet criteria for substance abuse or dependence in the past six months
* Female subjects will use barrier-method, non-hormonal contraception
* Capacity to understand all the relevant risks and potential benefits of the study (informed consent)
* Must be able to speak and read English

Exclusion Criteria:

* Current or past Axis I psychiatric diagnosis, including alcohol or substance abuse or dependence (except nicotine or caffeine), but not including minor Axis I disorders (e.g. simple phobia)
* Lifetime use of psychotropic medications, including antipsychotics, antidepressants, mood stabilizers, and anxiolytics
* Presence or history of medical or neurological illness that, in the judgment of the investigator, could influence the results of the study
* Diagnosis of diabetes, hemoglobin A1C > 6.5, hypertension, or dyslipidemias, or elevated random or fasting glucose, abnormal lipid levels, BP 130/85
* BMI 25 or < 19, history of BMI >35, and/or waist circumference >35 inches for females, 40 inches for males
* Subjects who are pregnant or breast-feeding or planning to become pregnant during the study
* Acute suicidality
* Meets criteria for a Diagnostic and Statistical Manual, Version 4 (DSM-IV) defined eating disorder
* Use of, or clinical indication for, one or more of the following medications: lithium, anti-epileptic medication, steroids (oral or inhaled), stimulants, serotonin reuptake inhibitors, mirtazapine, tricyclic antidepressants, thyroid supplementation, sibutramine, metformin, thiazolidinediones, beta-blockers, clonidine, niacin
* Subjects who have had >10% change in their body weight within the three months prior to enrollment
* HIV positive subjects
* Presence of mental retardation or pervasive developmental disorder
* History of recent (within 6 months) significant self-injurious behavior or violence
* Daily multivitamin or B-complex vitamin use
* A known history of dieting and difficulty with weight loss
* A strong family history of diabetes and/or heart disease
* History of congenital long QT syndrome or prolonged corrected QT interval (QTc) on screening EKG (>450ms)
* Concomitant use of any medication that inhibits 2D6 or 3A4 metabolism
* Low serum potassium or magnesium

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Ballon JS, Pajvani UB, Mayer LE, Freyberg Z, Freyberg R, Contreras I, Rosenbaum M, Leibel RL, Lieberman JA. Pathophysiology of drug induced weight and metabolic effects: findings from an RCT in healthy volunteers treated with olanzapine, iloperidone, or placebo. J Psychopharmacol. 2018 May;32(5):533-540. doi: 10.1177/0269881118754708. Epub 2018 Feb 15. PMID 29444618

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 69 consents in the study, 31 of which were randomized (started study medication). 24 subjects completed the study.
  The baseline characteristics reported were for the 24 subjects who completed the study.
Period: Overall Study
Arm/Group | Olanzapine | Iloperidone | Placebo
Started | 11 | 9 | 11
Completed | 7 | 7 | 10
Not Completed | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Iloperidone | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 10 | 24
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 6
  Male | 5 | 4 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 4 | 14
  White | 1 | 1 | 4 | 6
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 10 | 24
Starting BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.7 (0.3) | 23.6 (0.6) | 22.7 (0.5) | 23.0 (0.5)
Education (years) [Mean (Full Range); unit: years] | 16.4 [14 to 18] | 13.6 [12 to 16] | 14.9 [13 to 16] | 15 [12 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Delineate a pathophysiological mechanism of antipsychotic induced weight gain
Time Frame: baseline and 6 week visit
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
kg | 3.2 (1.0) | 0.8 (0.7) | 0.4 (0.5)

2. Primary Outcome: Change in Adiposity
Description: Total fat mass (excluding head) from baseline to Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
grams
  Baseline | 11942 (3635) | 14741 (7349) | 11690 (5469)
  Day 28 | 13312 (4246) | 16366 (6857) | 12081 (4649)

3. Secondary Outcome: Change in Leptin
Description: Leptin levels measured at Day 3 compared to baseline
Time Frame: change in baseline to Day 3
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
ng/dL | 2.47 (1.17) | 1.76 (0.8) | 1.16 (1.15)

4. Other Pre Specified Outcome: Change Glucose in People Taking Olanzapine or Iloperidone
Description: To quantify, prospectively, change in glucose from baseline to Day 28
Time Frame: Baseline to study termination (about 12 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
mg/dL
  Baseline | 11500.71 (2721.448) | 14430 (2148.776) | 10925.5 (1134.236)
  Day 28 | 11276.43 (1231.773) | 13975 (3813.754) | 12179.5 (1252.944)

5. Other Pre Specified Outcome: Change in Insulin
Description: Change in Insulin levels from baseline to Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: mlU/L
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
mlU/L
  Baseline | 9.7749 (3.42727) | 9.9316 (2.29266) | 10.9619 (2.66812)
  Day 28 | 12.0862 (7.39234) | 10.873 (5.9051) | 10.785 (2.62637)

6. Other Pre Specified Outcome: Insulin Resistance
Description: Homeostatic model assessment for Insulin Resistance (HOMA-IR) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
HOMA-IR score
  Baseline | 2.0477 (0.70188) | 2.0661 (0.56517) | 2.2988 (0.52346)
  Day 28 | 2.6147 (1.78901) | 2.4733 (1.60855) | 2.3362 (0.68093)

7. Other Pre Specified Outcome: Change in Food Intake
Description: Total grams of food consumed
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
grams
  Baseline | 1101.7715 (288.60787) | 1196.6557 (527.22574) | 1567.526 (608.53519)
  Day 28 | 1198.4071 (303.15123) | 1154.1286 (686.19597) | 1458.108 (731.06392)

8. Other Pre Specified Outcome: Change in Lipid Metabolism
Description: Change in lipid metabolism as measured by cholesterol/HDL ratio
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Olanzapine | Iloperidone | Placebo
Number analyzed (Participants) | 7 | 7 | 10
ratio
  Baseline | 2.71 (0.756) | 2.57 (0.787) | 2.7 (0.483)
  Day 28 | 3.14 (1.069) | 2.57 (0.787) | 2.5 (0.527)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Olanzapine | Iloperidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=7) | Iloperidone (N=7) | Placebo (N=10)
Drowsiness (General disorders) | 6 (6) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No